CLINICAL TRIAL: NCT03461523
Title: Observational, Prospective, Single-center Study: Should Body Mass Index (BMI) be Added to the Scoring Criteria of Hepatic Critically Ill Patients in Intensive Care Unit??
Status: Completed | Type: Observational
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Other Study IDs: BMI
Record Dates: First submitted 2018-03-03; First posted 2018-03-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: ICU Stay & Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to evaluate the hypothesis of poor clinical outcomes in critically ill patients that are having abnormal BMI.

DETAILED DESCRIPTION:
All demographic data will be obtained including the patients' age, sex, body mass index (BMI) & categorized into; BMI < 18.5Kg/m2 = underweight, BMI between 18.5-24.9Kg/m2 = normal weight, while BMI between 25-29.9Kg/m2 = overweight & obese = BMI ≥ 30Kg/m2, associated co-morbidities (diabetes mellitus, hypertension, chronic renal failure, cancer& chronic liver disease), the cause of admission to ICU, Sequential Organ Failure Assessment (SOFA), nutritional risk screening (NRS) on admission & discharge, prior cardiac arrest, previous ICU admission within 6months, nosocomial infection, organ failure e.g. cardiovascular, respiratory, renal & organic support requirement e.g. hemodynamic support, mechanical ventilation, renal replacement therapy (RRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the intensive care unit of National Hepatology & Tropical Medicine Research Institute (NHTMRI) for medical & surgical indications during the period from February 2018 to December 2020.

Exclusion Criteria:

* Patients will be excluded if they have stayed in ICU ≤24 hours and underweight (BMI<18.5).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that will be admitted to ICU will be categorized into; BMI < 18.5Kg/m2 =underweight, BMI between 18.5-24.9Kg/m2 = normal weight, while BMI between 25-29.9Kg/m2 = overweight & obese = BMI ≥ 30Kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
ICU stay | average 2 - 4 weeks
  Length of ICU stay in days
Mortality | average 2-4 weeks
  ICU Mortality in days

SECONDARY OUTCOMES:
the need for mechanical ventilation | during ICU stay 2-4 weeks
  notice & register the need for & type of mechanical ventilation; invasive or non invasive & days of ventilation
Duration of mechanical ventilation | 1-4 weeks
  Duration in days
the need for pharmacological support | 1-4 weeks
  notice & register the need for drugs to support the hemodynamics
occurrence of nosocomial infection | 2-28 days
  site of nosocomial infection
Hospital stay | average 2-28days
  Length of hospital stay
Hospital mortality | average 28 days
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt